CLINICAL TRIAL: NCT06263257
Title: The Effect of Mandala Art Therapy on Anxiety and Comfort Levels in Living Kidney Transplant Recipients: A Mixed-Methods Study
Brief Title: The Effect of Mandala Therapy on Anxiety and Comfort in Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Busra Nur Temur (Other)
Responsible Party: Sponsor-Investigator, Busra Nur Temur, Research Assistant, Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2023-631
Record Dates: First submitted 2024-01-18; First posted 2024-02-16 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-02

CONDITIONS: Anxiety; Transplant;Failure,Kidney; Transplant Complication
Keywords: kidney transplant; art therapy; anxiety; comfort; Randomized Controlled Trial
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Intervention group, the first measurement (afternoon of the day before surgery-T1) will include State-Trait Anxiety Inventory (STAI) and General Comfort Questionaire (GCQ), the second measurement (1 week after surgery-T2) will include State Anxiety Inventory and General Comfort Questionaire. The sessions of the Mandala Art Therapy training program for the intervention group will be conducted as follows: Session 1 on T2 (after the scales), Session 2 on 1st Control (2 week after surgery), Session 3 on 2nd Control (3 weeks after surgery-T3), and the third measurement at 3rd Control (3 weeks after surgery) (State Anxiety Inventory (STAI) and General Comfort Questionaire (GCQ).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Blinding In this study, blinding of participants and the statistician is planned. Blinding of the researcher implementing the intervention will not be possible. Since participants will not know to which group they are assigned, participant blinding is considered feasible. Data related to the scales (post-test) will be coded as 'A' and 'B' without indicating whether they belong to the intervention or control group. The coded data will be analyzed by a statistician, without knowledge of group allocation. After the statistical analyses are completed, the coding for the intervention and control groups will be revealed. This blinding technique is intended to minimize statistical bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): for the intervention group, the first measurement (afternoon of the day before surgery-T1) will include State-Trait Anxiety Inventory (STAI) and General Comfort Questionaire (GCQ), the second measurement (1 week after surgery-T2) will include State Anxiety Inventory and General Comfort Questionaire. The sessions of the Mandala Art Therapy training program for the intervention group will be conducted as follows: Session 1 on T2 (after the scales), Session 2 on 1st Control (2 week after surgery), Session 3 on 2nd Control (3 weeks after surgery-T3), and the third measurement at 3rd Control (3 weeks after surgery) will be collected through self-reporting for State Anxiety Inventory and General Comfort Questionaire.
  Interventions: Behavioral: Mandala Art Therapy
- Control Group (No Intervention): After obtaining consent from eligible participants within the scope of the study, the first measurement (STAI and GCQ) will be conducted on the afternoon of the preoperative day. Participants in this group will not be aware of their group assignment. The second measurement will be taken on postoperative day 5, the day of discharge (SAI and GCQ).
  The third measurement will be carried out during the participant's 3rd check-up after discharge (one month after surgery) for both STAI and GCQ. The intervention group's program will be shared with the control group participants on a voluntary basis after their discharge.

INTERVENTIONS:
Behavioral: Mandala Art Therapy — In art therapy, visual arts (such as drawing, painting, and sculpting) can be used as a tool to facilitate the expression of emotions and enhance coping skills. Naisin and colleagues (2006) reported that a one-hour art therapy session significantly reduced anxiety levels in hospitalized adult oncology patients. The word "mandala" is now typically associated with circular, geometric designs and often appears in adult coloring books aimed at promoting mindfulness and stress reduction. However, the methodology and theory of Jung related to mandalas are based not only on coloring pre-drawn templates but also on the activity of creating mandalas. The act of creating a mandala is claimed to provide immediate benefits in improving mood. The mandala is expressed as an instantaneous outward expression of the inner world of the person drawing it.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to evaluate the impact of mandala art therapy on the anxiety and comfort levels of living kidney transplant recipients. While kidney transplantation improves the recipients' quality of life, it may also expose them to psychological, physical, and social challenges post-transplant. This situation can increase recipients' levels of anxiety, making them cope with psychiatric issues and affecting their comfort levels. Feeling psychologically and physiologically comfortable is a crucial component of a successful recovery process for recipients.

Mandala art therapy is known as an effective method that supports the mental health, physical functioning, and social and emotional well-being of individuals with health issues. Mandalas can contribute to comfort by promoting inner peace, focusing attention, and encouraging creative expression. This study aims to investigate the impact of mandala art therapy on anxiety and comfort levels in kidney transplant recipients. To achieve this goal, a mixed-methods study using a randomized controlled and nested experimental design is planned.

The results of this study will provide valuable insights to healthcare providers by elucidating the impact of mandala art therapy on comfort and anxiety levels in living kidney transplant recipients. This information may guide healthcare professionals in enhancing kidney transplant recipients' psychological and emotional well-being, reducing stress, and promoting higher levels of comfort through mandala art therapy.

H0a: There is no effect of Mandala Art Therapy on the perceived anxiety level in living kidney transplant recipients.

H0b: There is no effect of Mandala Art Therapy on the comfort level of living kidney transplant recipients.

DETAILED DESCRIPTION:
This study is planned in three stages:

In the first stage, the preparation and pre-application of the Mandala Art Therapy training program for kidney transplant recipients in the intervention group will take place.

In the second stage, for the intervention group, the first measurement (afternoon of the day before surgery-T1) will include State-Trait Anxiety Inventory (STAI) and General Comfort Questionaire (GCQ), the second measurement (1 week after surgery-T2) will include State Anxiety Inventory and General Comfort Questionaire. The sessions of the Mandala Art Therapy training program for the intervention group will be conducted as follows: Session 1 on T2 (after the scales), Session 2 on 1st Control (2 week after surgery), Session 3 on 2nd Control (3 weeks after surgery-T3), and the third measurement at 3rd Control (3 weeks after surgery). For the Control Group, the third measurement (3 weeks after surgery) will be collected through self-reporting for State Anxiety Inventory and General Comfort Questionaire. This stage aims to conduct a randomized controlled study.

In the third stage, semi-structured interviews will be conducted with the intervention group, where the Mandala Art Therapy training program is implemented for kidney transplant recipients. Qualitative research methods will be employed in this stage (4 weeks after surgery).

The study population will consist of kidney transplant recipients admitted to the Organ Transplantation Clinic of Akdeniz University Hospital in Antalya, and those who apply to the Polyclinic of Prof. Dr. Tuncer Karpuzoğlu Organ Transplant Institute. In this center, 196 living donor kidney transplants were performed in 2021, 191 in 2022, and until June 19, 2023, 99 living donor kidney transplant surgeries have been carried out.

To enhance the robustness of the research findings and increase reliability, the study is planned to be conducted with a total of 72 participants, comprising 36 in the experimental group and 36 in the control group, representing a 40% increase during the course of the study.

Variables

Independent Variable:

Mandala Art Therapy Training

Dependent Variables:

State Anxiety Trait Anxiety Comfort Level

Randomization

In this study, random assignment and concealment of randomization are planned to control selection bias. Simple randomization will be used to allocate participants into the intervention and control groups. . The randomization process will be conducted by an individual who is not part of the research team. After the researcher confirms that the participant meets the inclusion criteria, does not meet any exclusion criteria, and obtains informed consent, the pre-test scales will be administered.

Blinding

In this study, blinding of participants and the statistician is planned. Blinding of the researcher implementing the intervention will not be possible. Since participants will not know to which group they are assigned, participant blinding is considered feasible. Data related to the scales (post-test) will be coded as 'A' and 'B' without indicating whether they belong to the intervention or control group. The coded data will be analyzed by a statistician, without knowledge of group allocation. After the statistical analyses are completed, the coding for the intervention and control groups will be revealed. This blinding technique is intended to minimize statistical bias.

State-Trait Anxiety Inventory (STAI)

The State-Trait Anxiety Inventory (STAI) was developed to assess state and trait anxiety in research and clinical applications. This scale consists of two subscales, State Anxiety and Trait Anxiety, each comprising 20 questions. Reliability and validity information for the STAI was reported in the psychometric information handbook by Spielberger. According to this report, Cronbach's Alpha (Internal Consistency) coefficient for the State Anxiety Scale is indicated as 0.73-0.86, and for the Trait Anxiety Scale, it is 0.86-0.93. The scale was adapted to Turkish and validated by Öner and Le Compte. The reliability of the scale was reported as Cronbach's Alpha coefficient of 0.83-0.92 for the State Anxiety Scale and 0.86-0.92 for the Trait Anxiety Scale.

The State Anxiety Scale describes how the individual feels in specific environmental conditions during a specific time interval when the test is administered. It is a Likert-type scale where a score between 1-4 can be given for each question. Participants are expected to mark only one of the options "1 (Not at all), 2 (Somewhat), 3 (Very much), 4 (Completely)" based on the intensity of their current feelings. The Trait Anxiety Scale requires participants to indicate how they mostly feel, marking one of the options "1 (Almost never), 2 (Sometimes), 3 (Often), 4 (Almost always)" based on the intensity of their feelings.

There are two types of expressions in the scales: direct expressions representing positive emotions and reversed expressions representing negative emotions. In the State Anxiety Scale, 10 items are reversed, and in the Trait Anxiety Scale, 7 items are reversed. When scoring reversed expressions, statements with a value of 1= are converted to 4= and those with a value of 4 are converted to 1. Scores obtained from both scales range between a minimum of 20 and a maximum of 80. A high score indicates a high level of anxiety, while a low score indicates a low level of anxiety. To calculate the State Anxiety and Trait Anxiety scores, the total score obtained for direct expressions is subtracted from the total score obtained for reversed expressions, and predetermined constant values are added. This value is 50 for the State Anxiety variable and 35 for the Trait Anxiety variable. The final value obtained represents the participant's anxiety score. A score of 0-19 indicates no anxiety, 20-39 indicates mild anxiety, 40-59 indicates moderate anxiety, and 60-79 indicates severe anxiety. An average anxiety score of 60 and above suggests that individuals need professional help. The Cronbach's alpha reliability coefficient will be calculated for the sample in this research. The permission letter for the "State-Trait Anxiety Inventory" was obtained on June 19, 2023, with the signature of Sibel Erenel, President of YÖRET Foundation, on behalf of Prof. Dr. Necla Öner.

General Comfort Questionnaire (GCQ)

The General Comfort Questionnaire, developed by Katharina Kolcaba, underwent a Turkish validation and reliability study conducted by Kuğuoğlu and Karabacak. (Cronbach's Alpha .85, .55-.85 for subscales). When testing the construct validity of the General Comfort Questionnaire and its sub-dimensions using the Satisfaction scale and its sub-dimensions, a significant positive relationship was found between the level of comfort and satisfaction with relaxation procedures (r=.225, p<0.05), satisfaction with nurses (r=.279, p<0.01), satisfaction with physicians (r=.199, p<0.01), satisfaction with auxiliary personnel (r=.198, p<0.01), satisfaction with meals (r=.206, p<0.01), satisfaction with the room (r=.214, p<0.01), and overall satisfaction with the hospital (r=.241, p<0.01). The scale consists of a total of 48 items and is presented in a four-point Likert type. The comfort levels of the scale are; relief (16 items), relaxation (17 items), and overcoming problems (15 items). The response orders of the scale, composed of positive and negative items, are given in a mixed manner. Accordingly, high scores (4) in positive items indicate high comfort and low scores indicate low comfort. In the evaluation of the scale, the obtained negative scores are reverse coded and summed with positive items. The highest total score that can be obtained from the scale is 192, and the lowest total score is 48. A low comfort score is expressed with one point, while a high comfort score is represented by four points. In Kolcaba's study, she determined Cronbach's alpha value for internal consistency control as .88 overall and as .66 - .80 for sub-scales. The Cronbach alpha reliability coefficient will be calculated for the sample of this study. The permission letter for the General Comfort Questionnaire was obtained on June 19, 2023, by Prof. Dr. Ükke Karabacak.

Data Analysis For the evaluation of the data obtained in the study, the IBM SPSS 23.0 software package will be utilized. Descriptive statistics will be presented using frequencies (n%) and mean±standard deviation (Min-Max) values. Pearson chi-square test and Fisher's Exact test will be employed for the analysis of relationships between categorical variables. The Shapiro-Wilks test will be used for the analysis of the normality assumption.

In cases where the assumption of the normal distribution is not met for the analysis of score differences between the two groups, the Mann-Whitney U test will be used when non-parametric, and the Student's t-test will be applied when parametric. For the non-parametric comparison of scores for three or more groups, the Kruskal-Wallis test will be utilized, and in cases where significance is found, the Bonferroni-Dunn test will serve as a post-hoc test. If the assumption of normal distribution is met, the ANOVA test will be employed for the comparison of scores for three or more groups, with the Tukey HSD test for pairwise comparisons.

For the analysis of the relationship between the scores of state and trait anxiety subscales and other variables, the Pearson correlation test will be conducted when the assumption of normal distribution is satisfied, and the Spearman correlation test will be used when it is not met. The Cronbach's alpha coefficient will be calculated for the reliability analysis of the scales.

A significance level of p<0.05 will be considered in the study.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Being a kidney transplant recipient
* Willing to participate voluntarily in the study
* Having person, place, and time orientation
* Undergoing kidney transplant for the first time

Exclusion Criteria:

* Having a diagnosed psychiatric illness
* Having a physical disability that would hinder drawing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Reduction in anxiety levels | First Measurement (Day Before Surgery): Second Measurement (Postoperative Day 5 - Discharge Day): Third Measurement (1 Month after Surgery - 3rd Control): The data will be reported six months after the completion of the data collection process.
  The first outcome is the change of continuous and situational anxiety levels in live kidney transplant recipients.
  The State-Trait Anxiety Inventory (STAI) was developed to assess state and trait anxiety in research and clinical applications. This scale consists of two subscales, State Anxiety and Trait Anxiety, each comprising 20 questions. Scores obtained from both scales range between a minimum of 20 and a maximum of 80. A high score indicates a high level of anxiety, while a low score indicates a low level of anxiety. This value is 50 for the State Anxiety variable and 35 for the Trait Anxiety variable. The final value obtained represents the participant's anxiety score. A score of 0-19 indicates no anxiety, 20-39 indicates mild anxiety, 40-59 indicates moderate anxiety, and 60-79 indicates severe anxiety. An average anxiety score of 60 and above suggests that individuals need professional help.
Increasing comfort level | First Measurement (Day Before Surgery): Second Measurement (Postoperative Day 5 - Discharge Day): Third Measurement (1 Month after Surgery - 3rd Control): The data will be reported six months after the completion of the data collection process.
  The second outcome is a change in the comfort levels of live kidney transplant recipients.
  General Comfort Questionnaire (GCQ) The scale consists of 48 items and is presented in a four-point Likert type. The comfort levels of the scale are; relief (16 items), relaxation (17 items), and overcoming problems (15 items). The response orders of the scale, composed of positive and negative items, are given in a mixed manner. Accordingly, high scores (4) in positive items indicate high comfort, and low scores (1) indicate low comfort. In the evaluation of the scale, the obtained negative scores are reverse coded and summed with positive items. The highest total score that can be obtained from the scale is 192, and the lowest total score is 48. A low comfort score is expressed with one point, while a high comfort score is represented by four points.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Nur Temür, M.Sc., Principal Investigator — Akdeniz University; Nilgün Aksoy, PhD, Study Director — Akdeniz University
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The sharing of all Individual Participant Data (IPD) underlying the results is planned
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD and any additional supporting information are planned to be shared in January 2025.
Access Criteria: The IPD and any additional supporting information will be shared with qualified researchers and analysts for specific types of analyses. Requests for access will be reviewed by Büşra Nur Temür based on established criteria, ensuring compliance with ethical and research guidelines

REFERENCES:
- [Background] Mantzios M, Giannou K. When Did Coloring Books Become Mindful? Exploring the Effectiveness of a Novel Method of Mindfulness-Guided Instructions for Coloring Books to Increase Mindfulness and Decrease Anxiety. Front Psychol. 2018 Jan 30;9:56. doi: 10.3389/fpsyg.2018.00056. eCollection 2018. PMID 29441038
- [Background] Abbing A, Ponstein A, van Hooren S, de Sonneville L, Swaab H, Baars E. The effectiveness of art therapy for anxiety in adults: A systematic review of randomised and non-randomised controlled trials. PLoS One. 2018 Dec 17;13(12):e0208716. doi: 10.1371/journal.pone.0208716. eCollection 2018. PMID 30557381
- [Background] Nainis N, Paice JA, Ratner J, Wirth JH, Lai J, Shott S. Relieving symptoms in cancer: innovative use of art therapy. J Pain Symptom Manage. 2006 Feb;31(2):162-9. doi: 10.1016/j.jpainsymman.2005.07.006. PMID 16488349